CLINICAL TRIAL: NCT02680522
Title: Study of Modulation Autonomic Heart Rate of Individuals With Parkinson's Disease and Healty Individuals Subject to a Training With Virtual Reality
Brief Title: Safety Study to Autonomic Rehabilitation o Parkinson's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Metodista de Piracicaba (Other)
Responsible Party: Principal Investigator, Rodrigo Santiago Barbosa Rocha, PhD student of the program in science of human movement, Universidade Metodista de Piracicaba
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 35683614.5.0000.5173
Record Dates: First submitted 2016-01-29; First posted 2016-02-11 (Estimated); Last update posted 2016-02-11 (Estimated); Status verified 2016-02

CONDITIONS: Parkinson Disease
Keywords: Parkinson's disease; Heart Rate Variability; Physiotherapy
MeSH Terms: conditions — Parkinson Disease | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control Group (Active Comparator): composed of healthy volunteers who underwent training with virtual reality. Exercises with game through virtual reality
  Interventions: Other: Exercise
- Parkinson's Group (Experimental): composed of patients with Parkinson's disease and who underwent training with virtual reality. exercises with game through virtual reality
  Interventions: Other: Exercise

INTERVENTIONS:
Other: Exercise — exercise training with virtual reality in videogame

SUMMARY:
Introduction: The Parkinson is one of the most common degenerative diseases of the central nervous system , mainly characterized by resting tremor , rigidity, akinesia and postural instability , also featuring the autonomic modulation of heart rate , which can lead to reduced frequency variability heart . Some activities may modify the modulation , including rehabilitation using virtual reality. Method: The research is interventional type , quantity and prospective, where volunteers were chosen for inclusion and exclusion criteria and divided into two groups , Control and Parkinson's, where they underwent 24 sections with virtual reality physiotherapy three times a week . Analysis of the autonomic modulation of heart rate was performed before and after the rehabilitation program with the frequency meter Polar brand. Statistical analysis was performed in 5.2 Biostat program with Shapiro- Wilk test to verify the normality , followed by t test to compare the data.

DETAILED DESCRIPTION:
To verify that the baseline conditions were adequate for the start of the collection, the volunteer remained 15 minutes at rest in supine position . They were measured and recorded : blood pressure by auscultation , using a mercury sphygmomanometer and a stethoscope ; and heart rate at rest by a heart rate monitor , with all measures carried out by the same researcher . Then the volunteer remained in the same position and was initiated to collect data with the registration of iR -R by Polar heart rate monitor model RS800CX (Polar Electro Co.Ltda . Kempele , Finland ) for 15 min. During the registration time, the participants maintained spontaneous respiration , were told not to talk , not sleep and avoid sudden movements . Subsequently , the recorded iR - R were transferred via an interface to a computer compatible for Polar softwere , the data being further processed into .txt format.

For the analysis we used the Kubius HRV Analysis Version 2.0 software (Kuopio, Finland). From the choice of the most stable stretch of five minutes, HRV was analyzed in the time domain (TD) and the variables selected the RR interval, the square root square mean difference between normal adjacent iR-R expressed in milliseconds (RMSSD) and SDNN, in the frequency domain via LF, HF and LF / HF addition to the non-linear analysis with the contents SD1, SD2 and Shannon Entropy.

To carry out the treatment with virtual reality Xbox 360® video game was the (Microsoft) used, the KinectTM Sensor, the kinectTM Adventures !, games with 6 modes and different phases and kinectTM Sports: Ultimate collection with 8 sports and different phases and TV Philips® the mark of 42 inches. The selected games were only the balance category, attention and planning, which consists of ten games, but only eight were used, including Kinect Sports game - "Tennis", "golf", "Ski" and the Kinect Adventure - "space bubble", "rapids", "top of the reflexes," "Hall of ricochets" and "leaks".

Before the first virtual training session , the presentation of the goals of each of the games and an adaptation session was held , where the therapists were next to the volunteer performing verbal commands . During the Games volunteers remained in the standing position and barefoot .

The volunteers performed 24 sessions in pairs, supervised by researchers for three times a week , every other day , lasting an hour each session. The scheduling range of care was organized so that the GP volunteers were always trained in the ON period of medication.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of Parkinson's Disease confirmed by medical evidence
* disease progression between three and ten years
* ranked between levels 2-3 in the modified Hoehn and Yahr
* with higher scores 24 or classified as illiterate score for the Mini-Mental State Examination.

Exclusion Criteria:

* With breathing problems induced by exercise
* orthopedic diseases
* with visual and / or hearing impairment
* uncontrolled hypertension
* use of vasoactive drugs
* which have performed heart surgery

Ages: 45 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Heart Rate Variability | evaluation before the beginning of the rehabilitation protocol and after 24 sessions (3 months)
  Data collection with the registration of iR-R by Polar heart rate monitor model RS800CX (Polar Electro Co.Ltda. Kempele, Finland) for 15 min. During the registration time, the participants maintained spontaneous respiration, were told not to talk, not sleep and avoid sudden movements. Subsequently, the recorded iR-R were transferred via an interface to a computer.
  For the analysis we used the Kubius HRV Analysis Version 2.0 software (Kuopio, Finland). 50 volunteers evaluation with Parkinson's disease and 50 healthy volunteers to investigate the improvement of autonomic modulation. all volunteers will be evaluated after three months of the end of the rehabilitation protocol in order to investigate whether the protocol improved the autonomic modulation in patients with Parkinson 's disease .

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Maués, Ms, Principal Investigator — Amazon University
Locations (1):
- Universidade da Amazônia, Belém, Pará, Brazil

IPD SHARING:
Plan to Share IPD: Yes
The data of the volunteers will be kept confidential , being only used the amount of data for publication in journals with the period until 2017

REFERENCES:
- [Result] Pompeu JE, Arduini LA, Botelho AR, Fonseca MB, Pompeu SM, Torriani-Pasin C, Deutsch JE. Feasibility, safety and outcomes of playing Kinect Adventures! for people with Parkinson's disease: a pilot study. Physiotherapy. 2014 Jun;100(2):162-8. doi: 10.1016/j.physio.2013.10.003. Epub 2013 Dec 27. PMID 24703891
- [Result] Montano N, Porta A, Cogliati C, Costantino G, Tobaldini E, Casali KR, Iellamo F. Heart rate variability explored in the frequency domain: a tool to investigate the link between heart and behavior. Neurosci Biobehav Rev. 2009 Feb;33(2):71-80. doi: 10.1016/j.neubiorev.2008.07.006. Epub 2008 Jul 30. PMID 18706440
- [Result] Broeren J, Claesson L, Goude D, Rydmark M, Sunnerhagen KS. Virtual rehabilitation in an activity centre for community-dwelling persons with stroke. The possibilities of 3-dimensional computer games. Cerebrovasc Dis. 2008;26(3):289-96. doi: 10.1159/000149576. Epub 2008 Jul 31. PMID 18667809
- [Result] Mihci E, Kardelen F, Dora B, Balkan S. Orthostatic heart rate variability analysis in idiopathic Parkinson's disease. Acta Neurol Scand. 2006 May;113(5):288-93. doi: 10.1111/j.1600-0404.2006.00580.x. PMID 16629763
- [Result] Saposnik G, Teasell R, Mamdani M, Hall J, McIlroy W, Cheung D, Thorpe KE, Cohen LG, Bayley M; Stroke Outcome Research Canada (SORCan) Working Group. Effectiveness of virtual reality using Wii gaming technology in stroke rehabilitation: a pilot randomized clinical trial and proof of principle. Stroke. 2010 Jul;41(7):1477-84. doi: 10.1161/STROKEAHA.110.584979. Epub 2010 May 27. PMID 20508185
- [Result] Haapaniemi TH, Pursiainen V, Korpelainen JT, Huikuri HV, Sotaniemi KA, Myllyla VV. Ambulatory ECG and analysis of heart rate variability in Parkinson's disease. J Neurol Neurosurg Psychiatry. 2001 Mar;70(3):305-10. doi: 10.1136/jnnp.70.3.305. PMID 11181850
- [Result] Vasilenko AF, Shamurov IuS, Mironova TF. [Sinus node activity in Parkinson's disease]. Klin Med (Mosk). 2011;89(3):47-50. Russian. PMID 21861404
- [Result] Niwa F, Kuriyama N, Nakagawa M, Imanishi J. Circadian rhythm of rest activity and autonomic nervous system activity at different stages in Parkinson's disease. Auton Neurosci. 2011 Dec 7;165(2):195-200. doi: 10.1016/j.autneu.2011.07.010. Epub 2011 Aug 25. PMID 21871844